CLINICAL TRIAL: NCT05846451
Title: Evaluating a Potential Pharmacokinetic Kratom-oxycodone Interaction Concurrent With Clinical Endpoints
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mary Paine, Professor, Washington State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19633; U54AT008909 (NIH)
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Herbal Interaction
Keywords: pharmacokinetic; pharmacokinetics; pharmacodynamic; pharmacodynamics; kratom; oxycodone; natural product; botanical product; natural product-drug interaction; mitragynine
MeSH Terms: interventions — mitragynine; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Sixteen non-naive* participants (8 males, 8 females) will be administered a single low dose (2 g) of a well-characterized kratom product by mouth as a tea. Pupil diameter will be measured from 0-12 hours. A washout of at least 10 days will separate Arms 1 and 2.
  *Non-naive subjects are defined as intermittent users who consume 2-8 g kratom at least once per month but no more than three times daily within the last six months prior to screening and are willing to abstain for several weeks
  Interventions: Dietary Supplement: Kratom
- Arm 2 (Active Comparator): The same 16 participants will be administered a single low dose (10 mg) of immediate-release oxycodone by mouth as a tablet. Plasma, pupil diameter measurements, and urine will be collected from 0-24 hours. A washout of at least 2 days will separate Arms 2 and 3.
  Interventions: Drug: Oxycodone
- Arm 3 (Experimental): The same 16 participants will be administered a single low dose (2 g) of kratom as a tea. After 15 minutes, the subjects will be administered a single low dose (10 mg) of oxycodone as a tablet by mouth. Plasma, pupil diameter measurements, and urine will be collected from 0-24 hours. A washout of at least 10 days will separate Arms 3 and 4.
  Interventions: Dietary Supplement: Kratom; Drug: Oxycodone
- Arm 4 (Experimental): The same 16 participants will self-administer a single low dose (2 g) of kratom as a tea once daily at home. On the fifth day, subjects will return to the research setting, where they will be administered a single low dose (2 g) of kratom, followed 15 minutes later by a single low dose (10 mg) of oxycodone by mouth. Plasma, pupil diameter measurements, and urine will be collected from 0-24 hours.
  Interventions: Dietary Supplement: Kratom; Drug: Oxycodone

INTERVENTIONS:
Dietary Supplement: Kratom — Kratom (Moon Kratom Yellow Indonesian, lot 51) is supplied as a dry leaf powder in clear plastic bags, each weighing 5 kg. Two grams of kratom dry leaf powder will be stirred into 240 mL of hot water to make a tea. The tea will be cooled to 50 degrees Celsius before administration. Participants will drink the tea within 15 minutes.
  Arms: Arm 1; Arm 3; Arm 4
Drug: Oxycodone — Immediate-release oral tablet, 10 mg
  Arms: Arm 2; Arm 3; Arm 4

SUMMARY:
The goal of this study is to investigate whether the botanical product kratom affects how the body processes the opioid drug oxycodone. The main research questions to be answered are two-fold:

1. How does kratom affect the manner in which oxycodone is metabolized (broken down and removed) by the body?
2. Does kratom change the effects oxycodone exerts on the body?

Healthy adult participants will complete four study arms, during which they will be given the following:

* Kratom (as a tea)
* A single dose of oxycodone (as a tablet)
* Kratom tea and a single dose of oxycodone
* Kratom tea for four days, then kratom tea and a single dose of oxycodone

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the potential for kratom to precipitate a pharmacokinetic interaction with the common opioid and dual cytochrome P450 (CYP) 3A/CYP2D6 substrate oxycodone. A secondary objective is to evaluate a potential pharmacodynamic interaction by measuring pupil diameter, the most sensitive measure of central nervous system opioid effects. To evaluate these objectives, participants will complete four arms, during which they will be administered the following:

* Arm 1: a single low dose of kratom (by mouth, as a tea)
* Arm 2: a single low dose of immediate-release oxycodone (by mouth, as a tablet)
* Arm 3: a single low dose of kratom tea and a single low dose of oxycodone
* Arm 4: daily at-home self-administration of kratom tea for four days, followed immediately by a single low dose of kratom tea and a single low dose of oxycodone in the research setting

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged from 21-45 years and healthy
* Body weight between 130 and 250 pounds (60-115 kg) and body mass index between 19 and 30
* Not taking any medications (prescription and non-prescription) or dietary supplements/botanical products known to alter the pharmacokinetics of either oxycodone or kratom
* Willing to abstain from consuming dietary supplements/botanical products and fruit juices for several weeks
* Willing to abstain from cannabis/marijuana, hemp, and THC- and/or CBD-containing products for several weeks
* Willing to abstain from consuming caffeinated beverages or other caffeine-containing products the evening before and morning of any inpatient visit
* Willing to abstain from consuming alcoholic beverages for one day prior to any inpatient visit
* Willing to use an additional method of contraception that does not include oral contraceptive pills, patches, or other hormonal methods (such as abstinence, copper IUD, or condoms)
* Have consumed kratom previously and tolerated it well without any unpleasant effects
* Willing to abstain from kratom for several weeks
* Have consumed any opioid previously and tolerated it well without any unpleasant effects or addiction
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for the subject to comply with the requirements of the study
* Geographically located within a 40-mile radius of Spokane and have the time to participate

Exclusion Criteria:

* Males and females under the age of 21 or over the age of 45
* People who weigh less than 130 pounds or more than 250 pounds
* People with a body mass index less than 19 or greater than 30
* Any current major illness or chronic illness including but not limited to kidney disease, hepatic disease, diabetes mellitus, hypertension, coronary artery disease, chronic obstructive pulmonary disease, cancer, or HIV/AIDS
* No previous exposure to kratom
* No previous exposure to an opioid
* History of anemia or any other significant hematologic disorder
* History of substance abuse, dependence, or addiction or major psychiatric illness
* A need for chronic opioid analgesics
* Use of opioid analgesics 3 weeks prior to initiation of the study
* An imminent likely need for opioid analgesics (e.g., planned dental or surgical procedure)
* Pregnant or nursing
* History of allergy or intolerance to kratom, other opioids, or oxycodone
* Taking concomitant medications, both prescription and non-prescription (including dietary supplements/botanical products), known to alter the pharmacokinetics of kratom or oxycodone
* Presence of a condition or abnormality that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data
* History of sleep apnea
* Any prior use of amphetamines, benzodiazepines, cocaine, MDMA, opioids, PCP, or other drugs for recreational purposes
* Use of cannabis/marijuana, hemp, THC-containing products, CBD-containing products, or CBD within the last month
* Out-of-range clinical laboratory value that the study physician considers participation in the study a health risk
* Inability to speak, read, and understand English

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Oxycodone area under the concentration vs. time curve (AUC) ratio (presence to absence of kratom) | 0-24 hours
  Ratio of the AUC of oxycodone in the presence to absence of kratom.

SECONDARY OUTCOMES:
Area under the pupil diameter (effect) vs. time curve (AUEC) ratio | 0-24 hours
  Ratio of AUEC in presence of oxycodone+kratom to oxycodone
Oxycodone maximum plasma concentration (Cmax) ratio (presence to absence of kratom) | 0-24 hours
  Ratio of Cmax of oxycodone in the presence to absence of kratom.
Oxycodone half-life ratio (presence to absence of kratom) | 0-24 hours
  Ratio of half-life of oxycodone in the presence to absence of kratom

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University College of Pharmacy and Pharmaceutical Sciences, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No